CLINICAL TRIAL: NCT02562118
Title: Phase Ib Followed by Phase II Study of Pre-operative Treatment With Lenvatinib Combined With Letrozole in Post-menopausal Women With Newly Diagnosed Hormone Receptor Positive Breast Cancer With Measurable Primary Breast Tumor
Brief Title: Neoadjuvant Lenvatinib Combined With Letrozole in Hormone Receptor Positive Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR01/04/15; 2015/00411 (Other: NHG DSRB)
Record Dates: First submitted 2015-09-08; First posted 2015-09-29 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: letrozole; lenvatinib
MeSH Terms: conditions — Breast Neoplasms | interventions — lenvatinib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenvatinib + Letrozole (Experimental): Single agent lenvatinib daily continuously x 2 weeks, followed by Letrozole 2.5mg daily + lenvatinib x 12 weeks (for Part A) or continuous till progression or intolerability (Part B)
  Interventions: Drug: Lenvatinib + Letrozole

INTERVENTIONS:
Drug: Lenvatinib + Letrozole — Single agent lenvatinib daily continuously x 2 weeks, followed by letrozole 2.5mg daily + lenvatinib x 12 weeks. Lumpectomy or mastectomy should be considered after completing 14 weeks of pre-operative lenvatinib + letrozole for curative intent in non-metastatic patients and for local control for patients with metastatic disease. If surgery is planned, it should preferably be performed within 2-12 weeks after completing neoadjuvant endocrine therapy, and after toxicities (if any) from the neoadjuvant endocrine therapy have resolved. If the patient is deemed inoperable after 14 weeks of lenvatinib + letrozole, a final biopsy will be obtained, and the patient discontinued from the study and treated as per standard clinical practice by the treating physician.

SUMMARY:
This is a single-centre study comprising two phases: a lead-in phase Ib and a phase II randomized portion.

Lead-in Phase Ib study A lead-in phase I study will be built into this protocol to confirm the dose of lenvatinib that can safely be combined with letrozole.

We expect that the optimal phase II dose level will be determined after recruiting 12-18 subjects into phase Ib. This dose level will be the one to be tested in the phase II portion of the study.

Phase II open label study In this part of the study, eligible patients will be treated with single agent lenvatinib at the phase II recommended dose for 2 weeks, followed by lenvatinib combined with letrozole 2.5mg daily for 12 weeks.

A total of 30 patients with ER positive breast cancer and measurable primary tumor will be enrolled over a period of 24-30 months

DETAILED DESCRIPTION:
Hypothesis:

We hypothesize that combining a RET inhibitor such as lenvatinib with endocrine therapy may potentiate anti-tumor effects in ER+ breast cancers in the clinic. Given that RET inhibition is the primary mechanism of action of lenvatinib, we further hypothesize that RET expression in the breast tumor may be a biomarker that predicts for better response to the combination of a RET inhibitor and endocrine therapy in both a neoadjuvant (Part A) and a metastatic (Part B) setting.

Primary Objectives

1. To confirm the dose of lenvatinib that can be safely combined with letrozole in the lead-in Phase Ib part of the study.
2. Part A (For patients with non-metastatic breast cancer undergoing neoadjuvant treatment) : To determine the overall clinical response (measured by ultrasound) and pathological complete response rate after 2 weeks of neoadjuvant single agent lenvatinib followed by 12 weeks of letrozole combined with lenvatinib and compare with historical controls treated with single agent letrozole.
3. Part B (For patients with metastatic breast cancer and who have tumor lesion that can be serially biopsied safely): to determine the clinical response (measured by RECIST criteria) after 2 weeks of single agent lenvatinib followed by continuous dual therapy of lenvatinib and letrozole, until time of progression or intolerability.

Secondary Objectives

1. To evaluate the overall biological effects (Ki67 changes, histological response, apoptosis, RET and downstream targets such as AKT and ERK) of 2 weeks of single agent lenvatinib, and of letrozole + lenvatinib, in ER positive breast cancer, respectively.
2. To identify biological predictors for treatment response to letrozole + lenvatinib in ER positive breast cancer using pharmacokinetics, pharmacogenetics, genomics and proteomics strategies.
3. To compare the following parameters between RET positive versus RET negative, ER positive breast cancer:

   * Part A :

i. Clinical response (measured by ultrasound) and biological effects of 2 weeks of single agent lenvatinib, ii. Clinical response (measured by ultrasound) and biological effects after 2 weeks of single agent lenvatinib followed by 12 weeks of letrozole combined with lenvatinib

-Part B : i. Clinical response measured by RECIST criteria after 2 weeks of single agent lenvatinib followed by letrozole combined with lenvatinib ii. Progression-free and overall survival with letrozole combined with lenvatinib

ELIGIBILITY:
Inclusion Criteria:

* Female, age ≥ 18 years.
* Histologic or cytologic diagnosis of breast carcinoma.
* Part A: T1-4 breast cancer with measurable primary breast tumor, defined as palpable tumor with both diameters 2.0cm or greater as measured by caliper. Newly diagnosed metastatic patients with measurable primary breast tumor ≥2cm are eligible provided that there are plans for toilet mastectomy after completing 14 weeks of pre-operative drug therapy. Patients must not have received prior chemotherapy or hormonal therapy for the treatment of the current breast cancer.
* Part B: Patients with metastatic breast cancer with measurable tumor by RECIST criteria.Patients previously treated with letrozole are eligible if they progressed on letrozole ≥1 year after adjuvant treatment, or ≥ 6 months in the metastatic setting.
* ECOG 0-1.
* Estimated life expectancy of at least 12 weeks.
* Adequate organ function including the following:

  * Bone marrow:
  * Absolute neutrophil (segmented and bands) count (ANC) ≥ 1.5 x 109/L
  * Platelets ≥ 100 x 109/L
  * Hepatic:
  * Bilirubin ≤ 1.5 x upper limit of normal (ULN),
  * ALT or AST ≤ 2.5x ULN, (or ≤5 X with liver metastases)
  * Renal:

Creatinine ≤ 1.5x ULN

• Post-menopausal women. Post-menopausal status is defined either by

* Age ≥ 60 years and one year or more of amenorrhea
* Age < 60 years and one year or more of amenorrhea (in the absence of ovarian suppression) and with estradiol and FSH levels consistent with menopause, *Treatment with a luteinizing hormone-releasing hormone (LHRH) agonist (goserelin acetate or leuprolide acetate) is not permitted for induction of ovarian suppression for Part A (patients with non-metastatic disease receiving the study treatment as neoadjuvant therapy).

However, in Part B (patients with metastatic disease), pre-menopausal women who are treated with medical ovarian suppression with post-menopausal levels of estradiol (institutional limits) at time of study entry and who will continue to be suppressed with 4-weekly LHRH agonist during study treatment may be enrolled. If these patients were previously on 12-weekly long-acting LHRH agonist, this has to be switched to 4-weekly LHRH agonist while the patient is on study treatment.

• Signed informed consent from patient or legal representative.

Exclusion Criteria:

* Treatment within the last 30 days with any investigational drug.
* Concurrent administration of any other tumor therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
* Major surgery within 28 days of study drug administration.
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Pregnancy.
* Breast feeding.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Active bleeding disorder or bleeding site.
* Non-healing wound.
* Poorly controlled diabetes mellitus.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Symptomatic brain metastasis.
* History of significant neurological or mental disorder, including seizures or dementia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-10-02 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Rates of clinical response | 2-3 weeks
  Complete and partial clinical response, including confidence intervals.

SECONDARY OUTCOMES:
Rates of pathological complete responses. | 4-6 weeks
  A pathological complete responder is defined as any patient who demonstrates no histological evidence of invasive tumor in the primary breast site as well as in resected axillary lymph nodes
Progression-free survival | 2 - 5 year
  Time to documented disease progression is defined as the time from the date of study enrollment to the first date of documented disease progression. Time to documented disease progression will be censored at the date of death for patients who have not had documented disease progression. For patients who are still alive at the time of analysis and who have not had documented disease progression, time to documented disease progression will be censored at the date of the last follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Lee, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Spanheimer PM, Park JM, Askeland RW, Kulak MV, Woodfield GW, De Andrade JP, Cyr AR, Sugg SL, Thomas A, Weigel RJ. Inhibition of RET increases the efficacy of antiestrogen and is a novel treatment strategy for luminal breast cancer. Clin Cancer Res. 2014 Apr 15;20(8):2115-25. doi: 10.1158/1078-0432.CCR-13-2221. Epub 2014 Feb 13. PMID 24526731
- [Background] Semiglazov VF, Semiglazov VV, Dashyan GA, Ziltsova EK, Ivanov VG, Bozhok AA, Melnikova OA, Paltuev RM, Kletzel A, Berstein LM. Phase 2 randomized trial of primary endocrine therapy versus chemotherapy in postmenopausal patients with estrogen receptor-positive breast cancer. Cancer. 2007 Jul 15;110(2):244-54. doi: 10.1002/cncr.22789. PMID 17538978